CLINICAL TRIAL: NCT04551313
Title: Effectiveness of Social Skills Training Group for Children With Autism Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202006158RINA
Record Dates: First submitted 2020-09-03; First posted 2020-09-16 (Actual); Last update posted 2023-08-18 (Actual); Status verified 2023-08

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism,autism spectrum disorder,social skill training
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- social skill training group (Experimental): We plan to address basic interactional and conversational skills first, then focus on teaching perspective-taking and theory of mind skills.
  Interventions: Behavioral: social skill group
- control group (Active Comparator): Regular therapy
  Interventions: Behavioral: social skill group

INTERVENTIONS:
Behavioral: social skill group — We plan to address basic interactional and conversational skills first, then focus on teaching perspective-taking and theory of mind skills.

SUMMARY:
Socio-communicative impairments are core deficits in individuals with autism spectrum disorder (ASD). Individuals with ASD have difficulty understanding eye contact, facial expressions, body language, and different tones of voice when communicating with others. They can't interpret the thoughts and feelings of others, or predict social events, and the impaired social skills may lead to rejection of peers and poor participation in school.

Social skills training targets the core symptoms of ASD. Empirical support is building for cognitive-behavioral intervention approach, social skills training group for verbally fluent, school-aged children with ASD. Several studies have shown the efficacy of the social story intervention. It is usually provided individually, but we want to use it in the group.

DETAILED DESCRIPTION:
Many different intervention program have been used throughout the world. One alternative method used to teach children is the social stories method, which was created by Gray (1993) to address the social difficulties of children with ASD. The theoretical framework of the social stories is based on theory of mind (TOM) hypothesis. Difficulties associated with the impaired TOM was addressed by explaining the complex social concepts in simple words and often include the description of perspectives of others. Several studies have shown the efficacy of the social story intervention. It is usually provided individually, but we want to use it in the group.

In this study, we plan to randomly assign thirty-six 5-7-year-old children with ASD to one of two kinds of social skills groups: the social skills group or the play activities group (control condition). Group met for 16 weeks, one time per week, one hour each time. Participants were recruited between October 2020 and September 2023. Assessment were conducted at baseline and endpoint (16 weeks). To empower parents, we would also ask parents of participants to attend our treatment and lecture.

ELIGIBILITY:
Inclusion criteria:

* Clinical diagnosis of Autism spectrum disorder
* Must be able to understand 3-steps verbal commands

Exclusion criteria:

* Mental retardation
* Seizure

Ages: 5 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2020-10-19 (Actual); Primary Completion 2022-07-27 (Actual); Study Completion 2022-07-27 (Actual)

PRIMARY OUTCOMES:
GAS (Goal attainment scale) | the first week and the 15th week of the duration
  interview caregivers about specific social interaction goals for the children and give rating 1-5 to calculate the extent to which a parent's goals are met.
Vineland Adaptive Behavior Scale | the first week and the 15th week of the duration
  to assess the socialization skill of the children.

CONTACTS AND LOCATIONS:
Overall Officials: Fu-Mei Chiang, MAMS, Principal Investigator — National Taiwan University Hospital
Locations (2):
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - NTUH, Taipei